CLINICAL TRIAL: NCT03682263
Title: Supported Employment Demonstration
Acronym: SED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: United States Social Security Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SS00-16-60014
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Mental Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Service Treatment (Experimental): The Full Service Arm receives the Individual Placement and Support (IPS) model of employment services integrated with behavioral health services and care management services, as well as Medication Management Support (MMS) from a Nurse Care Coordinator (NCC).
  Interventions: Behavioral: Full Service
- Basic Service Treatment (Experimental): The Basic Service Arm receives the Individual Placement and Support (IPS) model of employment services integrated with behavioral health services and care management services.
  Interventions: Behavioral: Basic Service
- Usual Services (No Intervention): Members of the Usual Service group seek services as they normally would (or would not) in their community. At the time of randomization, each Usual Services group member receives a comprehensive manual describing mental health and employment services in their local community, as well as state and national resources.

INTERVENTIONS:
Behavioral: Full Service — Receive Individual Placement and Support (IPS) model of employment services, behavioral health services, care management services, and Medication Management Support provided by a Nurse Care Coordinator (NCC).
  Arms: Full Service Treatment
Behavioral: Basic Service — Receive Individual Placement and Support (IPS) model of employment services, behavioral health services, and care management services.
  Arms: Basic Service Treatment

SUMMARY:
The purpose of this study is to determine whether offering an evidence-based package of employment supports integrated with mental health services has a positive impact on employment and clinical recovery, and delays or diminishes the need for disability benefits.

DETAILED DESCRIPTION:
SSA contracted with Westat to implement and evaluate the Supported Employment Demonstration (SED). The SED provides integrated mental health and vocational services to people with mental illness who were recently denied Social Security disability benefits. The evaluation will determine the impact of the SED on employment, clinical recovery, and receipt of disability payments. The evaluation is using a randomized controlled trial design to compare the outcomes of two treatment groups and a control group. In the full-service arm (n = 1,000), participants receive services from an Individual Placement and Support employment specialist, a care manager, and a nurse care coordinator (NCC) who provides medication management support, as well as modest funding for out-of-pocket prescriptions, essential work-related expenses, and other services in the participant's treatment plan. The basic-service arm (n=1,000), which is expected to cost about 50 percent less than the full-service arm, provides all services and funds except the NCC. Participants in the usual services (control) group (n = 1,000) seek services as they normally would but receive a comprehensive guide to local, state, and national resources.

Data collection includes computer-assisted baseline (in-person) and blinded quarterly (telephone) interviews with participants, collection of SSA administrative and site-level program data, site visits (including fidelity assessments), qualitative interviews with site administrators and service providers, focus groups with study participants, and person-centered ethnographic interviews with participants and nonparticipants.

ELIGIBILITY:
Inclusion Criteria:

* Individuals denied Social Security disability benefits (SSDI or SSI)
* Individuals alleging a mental impairment
* Live in Community Mental Health Agency (CMHA) catchment area
* Legally competent
* Express desire to improve work situation

Exclusion Criteria:

* Intellectual disability
* Reside in a nursing home or custodial institution
* Already receiving supported employment services from CMHA site

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Employment | 36 months
  Whether participant is employed in a paying job at any time during the 36 month study period.
  Assessed via quarterly computer-assisted telephone interviews.

SECONDARY OUTCOMES:
Employment (Competitive) | 36 months
  Whether a participant is employed in a community job that pays at least minimum wage (as defined by the resident state) and is "owned" by the employer rather than a mental health center or rehabilitation agency at any time during the 36 month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Total Hours Worked | 36 months
  The reported total number of hours worked for pay during the 36-month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Days to First Job | 36 months
  The number of days from enrollment date to first job during the 36-month study period, for those not employed at enrollment.
  Assessed via quarterly computer-assisted telephone interviews.
Months Employed | 36 months
  The number of months employed during the 36-month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Job Tenure | 36 months
  The longest number of consecutive months employed for any single job during the 36-month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Total Earnings | 36 months
  Total amount of reported earnings over the 36-month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Months above SGA | 36 months
  The number of months the participant reported earnings above Substantial Gainful Activity (SGA) levels over the 36-month study period.
  Assessed via quarterly computer-assisted telephone interviews.
Short-Form 12 Health Survey (SF-12) Mental Component Score (MCS) | 36 months
  The difference between the Short-Form 12 Health Survey (SF-12) Mental Component Score (MCS) measured at baseline (Baseline Survey) and at study exit (final quarterly follow-up survey).
  Higher values of the SF-12 MCS indicate better outcomes. A higher SF-12 MCS at study exit than at baseline indicates a positive change.
  Assessed via computer-assisted telephone interviews.
Time Until Award | 36 months
  The number of study days to disability award.
  Assessed using Social Security Administration administrative data.

CONTACTS AND LOCATIONS:
Overall Officials: William Frey, Ph.D., Principal Investigator — Westat; Robert Drake, MD, Ph.D., Principal Investigator — Westat
Locations (46):
- United States (46):
  - Penny Lane Centers, Lancaster, California
  - Mental Health Center of Denver, Denver, Colorado
  - Boley Centers, St. Petersburg, Florida
  - Trilogy, Chicago, Illinois
  - Bridgeway, Galesburg, Illinois
  - Bridgeway, Kewanee, Illinois
  - Bridgeway, Loves Park, Illinois
  - Bridgeway, Macomb, Illinois
  - Bridgeway, Normal, Illinois
  - Bridgeway, Pekin, Illinois
  - Mental Health Association of South Central Kansas, Wichita, Kansas
  - Communicare, Bardstown, Kentucky
  - Communicare, Brandenburg, Kentucky
  - Communicare, Elizabethtown, Kentucky
  - Communicare, Hardinsburg, Kentucky
  - Communicare, Hodgenville, Kentucky
  - Communicare, Lebanon, Kentucky
  - Communicare, Leitchfield, Kentucky
  - Communicare, Radcliff, Kentucky
  - Cornerstone Montgomery, Bethesda, Maryland
  - Pathways, Hollywood, Maryland
  - Cornerstone Montgomery, Rockville, Maryland
  - Cornerstone Montgomery, Silver Spring, Maryland
  - Pathways, Upper Marlboro, Maryland
  - Pathways, Waldorf, Maryland
  - Vinfen, Boston, Massachusetts
  - RISE, Minneapolis, Minnesota
  - Family Service League The Olsten Family Center, Bay Shore, New York
  - Family Service League The Olsten Family Center, East Hampton, New York
  - Family Service League The Olsten Family Center, Huntington, New York
  - Family Service League The Olsten Family Center, Mastic, New York
  - Family Service League The Olsten Family Center, Mattituck, New York
  - Greater Cincinnati Behavioral Health Services, Cincinnati, Ohio
  - The Nord Center, Lorain, Ohio
  - The Nord Center, Sheffield, Ohio
  - Mental Health Association Oklahoma, Tulsa, Oklahoma
  - Cascadia, Milwaukie, Oregon
  - Cascadia, Portland, Oregon
  - Anderson-Oconee-Pickens Mental Health Center, Anderson, South Carolina
  - Frontier Health, Bristol, Tennessee
  - Frontier Health, Greeneville, Tennessee
  - Frontier Health, Johnson City, Tennessee
  - Frontier Health, Kingsport, Tennessee
  - Helen Ross McNabb Center, Knoxville, Tennessee
  - Sunrise Services, Everett, Washington
  - Sunrise Services, Mount Vernon, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor JA, Salkever DS, Frey WD, Riley J, Marrow J. Enrollment in the Supported Employment Demonstration: An Employment Intervention for Denied Disability Benefits Applicants with a Mental Impairment. Adm Policy Ment Health. 2022 Nov;49(6):909-926. doi: 10.1007/s10488-021-01159-x. Epub 2021 Aug 17. PMID 34405312